CLINICAL TRIAL: NCT06302595
Title: Magnetic Resonance Imaging Guided Prostate Biopsy
Brief Title: MRI Guided Prostate Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Physical Sciences Inc. (Unknown)
Responsible Party: Principal Investigator, Kemal Tuncali, M.D., Assistant Professor of Radiology, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2022P001093; 5R44CA224853 (NIH)
Record Dates: First submitted 2024-02-15; First posted 2024-03-12 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Suspected Prostate Cancer
Keywords: prostate cancer; prostate biopsy; MR-guided prostate biopsy; targeted biopsy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MRI-guided prostate biopsy (Experimental): Participants who receive biopsy under MRI-guidance and a needle holder frame.
  Interventions: Device: MRI-guided prostate biopsy using the needle holder frame.

INTERVENTIONS:
Device: MRI-guided prostate biopsy using the needle holder frame. — A needle holding frame will be used during a routine MRI-guided prostate biopsy procedure, where tissue samples are obtained from each suspected region found on MRI using an MRI-conditional core biopsy needle. In this routine procedure, tissue sampling is performed in an MRI gantry and intraprocedural MRI is used to localize the regions.

SUMMARY:
This study aims to assess the feasibility of magnetic resonance (MR) guided prostate biopsy using a needle holder frame. This frame is used to help position the needle used for the biopsy. The feasibility in this study is defined as whether the needle holder frame enables accurate tissue sampling from a suspicious region in the prostate found on an MR image. If it does, a biopsy can be carried out with the needle holder frame safely in a clinical routine. The study will be conducted during a routine MR-guided prostate biopsy procedure with an investigational needle holder frame instead of a conventional needle-guiding template.

DETAILED DESCRIPTION:
The study will be conducted during a routine MR-guided prostate biopsy procedure. The following protocol follows the workflow of the routine procedure, except that the needle holder frame is used in place of a conventional needle-guiding template. The treating physicians have decided that an MR-guided prostate biopsy is necessary under the participant's current condition. If the participant chooses to participate in this research study, the procedure will be done in an MR scanner with an investigational needle holder frame.

Before the MR-guided prostate biopsy, the participant already had a standard clinical prostate MRI, the images from which will be used during the procedure.

The MR-guided prostate biopsy procedure may require monitored anesthesia or sedation. The participant will meet with the study physician prior to the biopsy procedure. The study physician will decide the type of monitored anesthesia or sedation to be used in discussion with the participant.

When undergoing a study in the MRI system, the participant will lie motionless inside the gantry of the system. Occasionally, the machine will produce a loud banging noise, as if it were being pounded from the outside with a hammer. Earplugs are available to reduce this sound level.

While the participant is in the magnet, under the anesthetic, the study physician will do the biopsy. To do this, the study physician will use a needle holder frame, which will show us where to put the needle by lining up the correct place outside on the skin or rectal wall.

Like the routine procedure, the biopsy is done with a needle put through the skin under the participant's scrotum by the doctor. The location of the needle is confirmed by acquiring an MR image (confirmation image). Several biopsies are taken each time, from either side of the gland and from places where the MR images show shadows or abnormal areas. There can be a range of 6-15 locations to sample. Because the location of the needle is always confirmed on the confirmation image, like the routine procedure, the use of the needle holder frame will not compromise the sampling of MR-indicated abnormal areas. The participant will be in the study for about 1.5 hours, which is how long the biopsy procedure will take. After the procedure, the investigator will review the confirmation images to assess the accuracy of needle placement, though it will not change the health outcome (e.g., pathological findings).

ELIGIBILITY:
Inclusion Criteria:

* Either an abnormal serum prostate-specific antigen (PSA) level (> 4ng/Ml) or a palpable nodule in the prostate on digital rectal examination or prostate MRI suspicious lesion..
* Diagnostic MRI of the prostate gland.
* Age > 30 years
* Signed informed consent.
* No contra-indications to MRI, i.e. no cardiac pacemaker.
* No recent or ongoing active ischemic heart disease.

Exclusion Criteria:

* Inability to give informed consent.
* Contra-indications to MRI- cardiac pacemaker, inner ear implants, non-MR compatible intracranial aneurysm clips.
* Recent or ongoing active ischemic heart disease such as recent or ongoing angina.

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of needle placement | During the MRI-guided prostate biopsy procedure
  The number of biopsy failures (defined as the number of needle insertions that miss the target zone defined on MRI).

CONTACTS AND LOCATIONS:
Overall Officials: Kemal Tuncali, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No